CLINICAL TRIAL: NCT06685653
Title: An Exploratory Study of Personalized Neoantigen MRNA Vaccine RGL-270 Combined with Adebrelimab in Non-Small Cell Lung Cancer Patients
Brief Title: Personalized Neoantigen MRNA Vaccine Combined with Adebrelimab in Non-Small Cell Lung Cancer Patients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanjing Tianyinshan Hospital (Other)
Collaborators: Jilin Provincial Cancer Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-IIT-RGL-270-TYS
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: NSCLC
Keywords: NSCLC; Personalized mRNA tumor vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: Resectable NSCLC subjects (Experimental)
  Interventions: Biological: Adebrelimab+RGL-270
- Part B: NSCLC subjects with disease recurrence or metastasis after first-line standard therapy (Experimental)
  Interventions: Biological: Adebrelimab+RGL-270/single RGL-270

INTERVENTIONS:
Biological: Adebrelimab+RGL-270 — Drug: Adebrelimab Adebrelimab is a programmed death-ligand 1 antibody.
  Drug: RGL-270 RGL-270 is a mRNA tumor vaccines
  Arms: Part A: Resectable NSCLC subjects
Biological: Adebrelimab+RGL-270/single RGL-270 — Drug: Adebrelimab Adebrelimab is a programmed death-ligand 1 antibody.
  Drug: RGL-270 RGL-270 is a mRNA tumor vaccines
  Arms: Part B: NSCLC subjects with disease recurrence or metastasis after first-line standard therapy

SUMMARY:
This is a phase IIT , it is an open-label study designed to evaluate the safety and tolerability of personalized mRNA tumor vaccine RGL-270 targeting tumor-specific neoantigens and Adebrelimab (a humanized PD-L1 monoclonal antibody) in patients with resectable NSCLC and those with NSCLC who have relapsed or metastasized after first-line standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Part A & Part B

  1. Subjects should understand and comply with the relevant procedures of the study, and voluntarily sign the pre-screening informed consent form;
  2. Age 18-75 years old (including boundary value), gender is not limited;
  3. Willing to provide tumor tissue specimens for genetic testing and neoantigen analysis;
  4. United States Eastern Cooperative Oncology Group (ECOG) score: 0 or 1 point;
  5. Estimated survival ≥ 6 months;
  6. Willing to provide blood samples required for the detection of immunogenicity and biomarkers before and after treatment, of which the blood samples for genetic testing during the screening period must be free of blood transfusions, blood products and other hematopoietic stimulating factors within 7 days before collection;
  7. Vital organ function meets the following criteria (no use of any blood components and cell growth factors within 14 days prior to initiation of study treatment):

     ① Routine blood count: neutrophil count (ANC) ≥ 1.5×109/L, lymphocyte count (LYM) ≥0.5×109/L, platelet count (PLT) ≥1× lower limit of normal (LLN), hemoglobin (Hb) ≥90g/L;

     ② Blood biochemistry: total bilirubin (TBIL) ≤ 1.5× upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5× ULN, serum albumin (ALB) ≥30g/L, serum creatinine (Scr) ≤ 1×ULN;

     ③ Coagulation routine: international normalized ratio (INR) ≤ 1.5, activated partial thromboplastin time (APTT) ≤ 1.5×ULN;

     ④ Cardiac function: left ventricular ejection fraction (LVEF) ≥50%;

     ⑤ ECG: Fridericia's corrected QT interval (QTcF) <470 msec; The QTc interval must be corrected according to Fridericia's criteria by the formula QTcF = QT/RR^0.33.
  8. Female subjects of childbearing potential must have a serum pregnancy test within 7 days prior to the first dose with a negative result; and must be non-lactating;
  9. Female subjects of childbearing potential and male subjects whose partners are women of childbearing potential must agree to comply with contraceptive requirements from the time of signing the informed consent form until 90 days after the end of the last treatment session (see "Contraceptive Methods" in Annex V for details).

     Part A
  10. Surgically resected stage IIB, IIIA, STAGE IIIB (N2) NSCLC with histologically or cytologically confirmed according to United States Joint Committee on Cancer (AJCC) 8th edition guidelines;
  11. Received 3-4 cycles of neoadjuvant therapy with platinum-containing doublet combined with immune checkpoint inhibitors, and the tumor histopathology showed that the main pathological response (MPR) was not achieved after radical resection (R0 resection); No neoadjuvant therapy requiring surgery to achieve R0 resection; (Note: Major pathologic response (MPR) is defined as the percentage of residual viable tumor cells in the tumor bed after neoadjuvant therapy ≤ 10%, regardless of whether there are viable tumor cells remaining in the lymph nodes.) ）
  12. Postoperative complications have recovered, or complications are lower than Clavien-Dindo complication grade 3;
  13. There was no evidence of disease on clinical examination, baseline radiological assessment of chest and abdomen CT and head MRI within 14 days prior to the first dose of vaccine.

      Part B
  14. Histologically or cytologically confirmed locally advanced unresectable or recurrent/metastatic NSCLC;
  15. Disease progression during or after first-line platinum-containing therapy (with or without immunotherapy);
  16. At least one measurable solid tumor lesion according to RECIST 1.1 criteria. (Note: Lesions that have received prior radiotherapy should not be used for target lesions unless there is clear radiographic progression after radiotherapy.) ）

Exclusion Criteria:

Part A & Part B

1. Histologically or cytologically confirmed small cell carcinoma (SCLC), mixed SCLC and NSCLC, or other non-NSCLC;
2. Carriers of driver mutations (including but not limited to EGFR and ALK gene alterations) for which targeted drugs have been approved for marketing and are accessible;
3. Received immune cell or tumor vaccine treatment, including but not limited to tumor-infiltrating lymphocytes (TILs), chimeric antigen receptor T cells (CAR-T), T cell receptor chimeric T cells (TCR-T), and therapeutic tumor vaccines;
4. Administration of live attenuated vaccine within 28 days prior to the screening period or planned administration during the study and within 90 days after the end of study drug treatment (inactivated vaccine is allowed);
5. Any person who is not suitable for immunotherapy as assessed by the investigator;
6. Presence of autoimmune diseases, except for hypothyroidism requiring hormone replacement therapy due to autoimmune thyroiditis;
7. Evidence of active tuberculosis infection within 1 year prior to the screening period, regardless of treatment;
8. Subjects with a known history of interstitial pneumonia or a high suspicion of interstitial pneumonia, or evidence of active interstitial pneumonia on chest CT during the screening period; Known history of idiopathic pulmonary fibrosis, history of organizing pneumonia (e.g., bronchiolitis obliterans or cryptogenic organizing pneumonia);
9. Concurrent severe infection within 28 days prior to the screening period (such as the need for intravenous infusion of antibiotics, antifungal or antiviral drugs according to clinical diagnosis and treatment standards), or the presence of active infection requiring intravenous infusion of antibiotics during the screening period;
10. Presence of clinically uncontrolled pleural effusion or ascites requiring thoracentesis or paracentesis drainage within 14 days prior to the screening period;
11. Known allergy to the study drug or any of its excipients, or history of severe allergic reactions to other vaccines;
12. History of other malignancies within the past 5 years, excluding cured carcinoma in situ of the cervix, basal cell carcinoma of the skin or squamous cell carcinoma of the skin, localized prostate cancer after radical resection, ductal carcinoma in situ after radical resection (hormonal therapy for non-metastatic prostate cancer or breast cancer is allowed), and papillary thyroid carcinoma;
13. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
14. Patients with congenital or acquired immunodeficiencies, such as cellular immunodeficiencies (e.g., DiGeorge syndrome, T-negative severe combined immunodeficiency [SSCID]) or combined T-cell and B-cell immunodeficiencies (e.g., T- and B-negative combined immunodeficiency, Wiskott-Aldrich syndrome, ataxia telangiectasia, common variable immunodeficiency); or human immunodeficiency virus (HIV) infection;
15. Active hepatitis B (defined as a positive test result for active hepatitis B virus surface antigen [HBsAg] at the screening period with detection of HBV DNA ≥500 IU/mL or above the upper limit of normal testing at the research center), or hepatitis C (defined as a positive test result for hepatitis C antibody [HCV-Ab] and positive HCV-RNA during the screening period);
16. Has poorly controlled or severe cardiovascular disease: if there is symptomatic congestive heart failure (NYHA class III. or IV.), or myocardial infarction within 6 months prior to the screening period, or unstable angina within 1 month prior to the screening period, or there is a severe cardiac arrhythmia requiring treatment or intervention, or there is hypertension (systolic blood pressure ≥ 160mmHg, diastolic blood pressure ≥ 100mmHg that is still poorly controlled after adequate treatment);
17. Other circumstances that may affect the conduct of the clinical study and the judgment of the results of the study as judged by the investigator (such as the subject's possible poor compliance, or any other disease that puts the subject at risk to safety, or the analysis results of tumor tissue sequencing data show that there is not enough neoantigen available for vaccine preparation, or the vaccine preparation fails).

    Part B
18. Has active leptomeningeal disease or uncontrolled and untreated brain metastases;
19. Toxicity from prior antineoplastic therapy has not recovered to baseline or ≤ grade 1 (except for alopecia and pigmentation), and neurotoxicity has not recovered to grade ≤2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Primary Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
• Incidence of DLTs | 21 days after first administration of RGL-270 in combination with Adebrelimab
  • Incidence of DLTs during the observation period of dose-limiting toxicities (DLTs).
• Safety endpoints | 90 days (± 7 days) after the last vaccine/adebelimab treatment or 30 days (±7 days) after the last chemotherapy
  laboratory indicators, 12-lead ECG, United States Eastern Cooperative Oncology Group (ECOG) performance status score, physical examination, vital signs, adverse events/serious adverse events (AEs/SAEs, severity according to NCI-CTCAE v5.0 criteria)

SECONDARY OUTCOMES:
Change from baseline of LNPs | 18 months/24 months after the first dose
  To evaluate the changes of nanolipid particles (LNPs) in peripheral blood after administration
Change from baseline of neoantigen-specific T cell | 18 months/24 months after the frst dose
  Change from baseline in neoantigen-specific T cell response positivity rate and response signaling
Change from baseline of ADA | 18 months/24 months after the frst dose
  Change from baseline in anti-personalized tumor vaccine RGL-270 and/or adebelimab anti-drug antibody (ADA)
The DFS, OS, DFS rate and OS rate in Resectable NSCLC | 18 months/24 months after the frst dose
  Resectable NSCLC: disease-free survival (DFS), overall survival (OS), DFS rate at 18 months/24 months post-dose, and OS rate
The ORR, DoR, PFS and OS in Advanced NSCLC | 18 months/24 months after the frst dose
  Advanced NSCLC: objective response rate (ORR), duration of response (DoR), progression-free survival (PFS), OSTime Frame: 18 months/24 months after the first dose